CLINICAL TRIAL: NCT05120297
Title: A Study to Evaluate the Efficacy and Safety of AK101 in Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: A Phase 3 Study of Efficacy and Safety of AK101 in Subjects With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK101-302
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK101 (Experimental)
  Interventions: Drug: AK101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK101 — Subjects will receive AK101 subcutaneous injection at week 0 and week 4, and will follow up to week 16.
  Arms: AK101
Drug: Placebo — Subjects will receive placebo subcutaneous injection at week 0 and week 4, and will follow up to week 16.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicentered phase III clinical study to evaluate the efficacy and safety of AK101 in the treatment of subjects with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter phase III clinical study. The purpose of this study is to evaluate the efficacy and safety of AK101 in the treatment of subjects with moderate-to- severe plaque psoriasis. Subjects will be randomized to receive AK101 or placebo injection subcutaneously, and follow up to week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years.
2. Subjects diagnosed with moderate-to-severe plaque psoriasis for at least 6 months before screening.
3. At screening and baseline, PASI score ≥ 12, Body Surface Area BSA (BSA) ≥ 10%, sPGA ≥ 3.
4. Subjects with a history of an inadequate response, intolerable or medically inappropriate use of systemic therapy and/or phototherapy.
5. Subjects who are women of childbearing potential must have a negative pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 6 months after the last study drug administration.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type psoriasis.
2. History or evidence of active TB. Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment had initiated and maintained according to protocol.
3. Positive results of confirmatory test for hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or syphilis.
4. History of repeated chronic infection, had any serious infection or systemic infection within 2 months before screening.
5. History of prohibited psoriasis treatments within 2/4 weeks before randomization.
6. History of IL12/23 or IL-23 inhibitors therapy.
7. Inadequate washout period of prior biological therapy.
8. History of malignant tumour within 5 years before screening.
9. Any medical or psychiatric condition, laboratory, or ECG parameter which, in the opinion of the Investigator would place the subject at risk, interfere with participation or interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who achieved at least 75% (PASI 75) reduction in psoriasis area and severity index (PASI) score from baseline. | At week 16
Percentage of subjects who achieved static physician global assessment (sPGA) clearance or very slight (0/1). | At week 16

SECONDARY OUTCOMES:
Percentage of subjects who achieved at least 50% (PASI 50), 75% (PASI75, except week 16) and 90% (PASI 90) reduction in PASI score at each visit. | Baseline to week 16
Percentage of subjects who achieved sPGA 0/1 at each visit. | Baseline to week 16
Percentage change of PASI from baseline. | Baseline to week 16
PK: AK101 serum concentration at different time points after administration. | Baseline to week 16
Immunogenicity assessment: number and percentage of subjects with detectable anti-AK101 antibody (ADA). | Baseline to week 16
Safety: Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAE). | Baseline to week 16

CONTACTS AND LOCATIONS:
Locations (52):
- China (52):
  - AkesoBio Investigative Site 1010, Bengbu, Anhui
  - AkesoBio Investigative Site 1028, Hefei, Anhui
  - AkesoBio Investigative Site 1013, Wuhu, Anhui
  - AkesoBio Investigative Site 1001, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1027, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1034, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1035, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1036, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1049, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1051, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1041, Chongqing, Chongqing Municipality
  - AkesoBio Investigative Site 1007, Guangzhou, Guangdong
  - AkesoBio Investigative Site 1021, Guangzhou, Guangdong
  - AkesoBio Investigative Site 1024, Guangzhou, Guangdong
  - AkesoBio Investigative Site 1018, Shenzhen, Guangdong
  - AkesoBio Investigative Site 1023, Shenzhen, Guangdong
  - AkesoBio Investigative Site 1030, Shenzhen, Guangdong
  - AkesoBio Investigative Site 1012, Nanning, Guangxi
  - AkesoBio Investigative Site 1039, Guiyang, Guizhou
  - AkesoBio Investigative Site 1025, Chengde, Hebei
  - AkesoBio Investigative Site 1017, Shijiazhuang, Hebei
  - AkesoBio Investigative Site 1031, Shijiazhuang, Hebei
  - AkesoBio Investigative Site 1014, Harbin, Heilongjiang
  - AkesoBio Investigative Site 1033, Nanyang, Henan
  - AkesoBio Investigative Site 1045, Zhengzhou, Henan
  - AkesoBio Investigative Site 1004, Wuhan, Hubei
  - AkesoBio Investigative Site 1006, Changsha, Hunan
  - AkesoBio Investigative Site 1026, Changsha, Hunan
  - AkesoBio Investigative Site 1052, Lianyungang, Jiangsu
  - AkesoBio Investigative Site 1029, Nanjing, Jiangsu
  - AkesoBio Investigative Site 1009, Xuzhou, Jiangsu
  - AkesoBio Investigative Site 1015, Yancheng, Jiangsu
  - AkesoBio Investigative Site 1019, Nanchang, Jiangxi
  - AkesoBio Investigative Site 1020, Nanchang, Jiangxi
  - AkesoBio Investigative Site 1032, Changchun, Jilin
  - AkesoBio Investigative Site 1047, Changchun, Jilin
  - AkesoBio Investigative Site 1008, Dalian, Liaoning
  - AkesoBio Investigative Site 1048, Shenyang, Liaoning
  - AkesoBio Investigative Site 1050, Hohhot, Neimenggu
  - AkesoBio Investigative Site 1044, Yinchuan, Ningxia
  - AkesoBio Investigative Site 1038, Jinan, Shandong
  - AkesoBio Investigative Site 1042, Jinan, Shandong
  - AkesoBio Investigative Site 1043, Qingdao, Shandong
  - AkesoBio Investigative Site 1005, Shanghai, Shanghai Municipality
  - AkesoBio Investigative Site 1046, Taiyuan, Shanxi
  - AkesoBio Investigative Site 1011, Chengdu, Sichuan
  - AkesoBio Investigative Site 1016, Suining, Sichuan
  - AkesoBio Investigative Site 1040, Tianjin, Tianjin Municipality
  - AkesoBio Investigative Site 1037, Kunming, Yunnan
  - AkesoBio Investigative Site 1002, Hangzhou, Zhejiang
  - AkesoBio Investigative Site 1003, Hangzhou, Zhejiang
  - AkesoBio Investigative Site 1022, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No